CLINICAL TRIAL: NCT01523561
Title: Influencing Adolescent Girls With Internalizing Problems With Creative Dance Twice Weekly. A Randomised, Controlled Study
Brief Title: Influencing Adolescent Girls´ With Creative Dance Twice Weekly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Margareta Moller, professor, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMO027
Record Dates: First submitted 2012-01-18; First posted 2012-02-01 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Adolescent - Emotional Problem
Keywords: dance; intervention; adolescent; girls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): The participants in the no intervention group were informed that they should continue living as usual
- dance intervention (Experimental): The dance intervention took place twice weekly for a period of 1 year under the guidance of two dance class teachers. The duration of the class was 75 min. and the dance training was always carried out to popular music. The dance choreography was adjusted to the level of the participants' skills in order to make them feel successful in their exercise. During the intervention year, the theme of dance styles varied from hip hop, jazz and contemporary dance. African dance was used in the warm up section. The dance class always ended with a relaxation. The dance intervention had a focus on emphasizing the participants' resources and creates a feeling of affinity. Listening to signals from the body, reducing focus on the performance and "become part of the movement" was encouraged.
  Interventions: Behavioral: dance group

INTERVENTIONS:
Behavioral: dance group — The dance intervention took place twice weekly for a period of 1 year under the guidance of two dance class teachers. The duration of the class was 75 min. and the dance training was always carried out to popular music. The dance choreography was adjusted to the level of the participants' skills in order to make them feel successful in their exercise. During the intervention year, the theme of dance styles varied from hip hop, jazz and contemporary dance. African dance was used in the warm up section. The dance class always ended with a relaxation. The dance intervention had a focus on emphasizing the participants' resources and creates a feeling of affinity. Listening to signals from the body, reducing focus on the performance and "become part of the movement" was encouraged.
  Arms: dance intervention

SUMMARY:
The aim of this study is to evaluate if creative dance twice weekly can influence girls wellbeing. The focus lies on girls 13-18 years old that suffer from repeatedly psychosomatic problems and/or stress.

Specific objectives are

* To assess the effect of the dance intervention in reducing psychosomatic problems (such as pain in the head, neck, shoulder or stomach), stress and depression
* Determine which factors are important for continuing dancing and keeping up new habits
* A cost-effectiveness analyse of the health outcome.

Geographical area: Örebro County (population 276,000)

DETAILED DESCRIPTION:
The school nurses asked girls aged 13-18 years old, who searched for psychosomatic problems, if they wished to participate in the dance project. Recruitment of girls where also carried out in information about the project at parent meetings and in school classrooms. 143 girls completed the base-line questionnaire, 138 met the inclusion criteria and were included. Randomization was carried out to intervention and control group.

The quantitative data collection is carried out with a questionnaire. Participants in the dance intervention and the control group will response to this questionnaire at 7 times during the study, at start and every six months over a total period of 3 years.

Girls who are found to be at risk of having severe depression (> 34 points) in the depression scale CES-DC met with an experienced licensed psychologist. This was to explore if there was a need for extended support and help and the girl's parents and Child and Adolescent Psychiatric Care was contacted in most cases and if there was a risk for suicide. The results from the depression scale at base - line (CES-DC) showed that 81% of the girls in the study had depressive symptoms and 29% had high levels of depressive symptoms.

The qualitative interviews were performed in order to explore the girls experience of the dance lessons and to assess if and/or how dance intervention has affected her self-esteem in any way. These interviews were conducted on a strategic sample of 20 girls who participated in the dance intervention.

The dance intervention took place in a gym in Örebro twice weekly for a period of 1 year under the guidance of two dance class teachers (one at a time). The duration of the class was 75 minutes and the dance training was always carried out to popular and suitable music. The dance choreography was adjusted to the level of the participants' skills in order to make them feel successful in their exercise. During the intervention year, the theme of dance styles varied from hip hop, jazz, aerobic dance and contemporary dance. African dance, to the music of African drums, was used in the warm up section. The dance class always ended with a 10-min-relaxation training. The dance intervention had a strong focus on emphasizing the participants' resources and creates a feeling of affinity. The dance teachers encouraged them to listen to signals from the body, reducing focus on the performance and "become part of the movement".

ELIGIBILITY:
Inclusion Criteria:

* The study population comprised adolescent girls with internalizing problems who had recurrent visits to the school nurse due to psychosomatic symptoms such as:

  * pain in the head, stomach, neck, back and/or shoulder.
  * persistent feelings of tiredness
  * being worried
  * in low spirit or depressed were also inclusion criteria.

Exclusion Criteria:

* severe hearing impairment
* intellectual disability
* difficulties with the Swedish language or
* if the CAP had advised against participation.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Self reported health | change from baseline to follow up at 20 months
  the single-item question "How do you rate your general health?" is frequently used in national and international surveys. The response alternatives is 1. Very poor, 2. Poor, 3. Neither good nor poor, 4. Good, 5. Very good. Measuring general health with a five-degree scale has been agreed upon in the EU.

SECONDARY OUTCOMES:
adherence to and experience of the intervention | change baseline to follow up at 20 months
  The adherence to the dance intervention was measured by registering attendance at every dance session during the intervention period. Cancellations were made by telephone or text message.The experience of the dance intervention was evaluated with a graphic rating scale, a modified Visual Analogue Scale with five discrete alternatives.The question was "How do you experience dancing while you perform it?"; the rating scale started at "entirely negative" and ended at "entirely positive." Cut-off was set between "neutral" and "entirely positive".

CONTACTS AND LOCATIONS:
Overall Officials: Margareta HL Moller, professor, Principal Investigator — Örebro County Council
Locations (1):
- Centre for health care Sciences, Örebro, Närke, Sweden

REFERENCES:
- [Derived] Philipsson A, Duberg A, Moller M, Hagberg L. Cost-utility analysis of a dance intervention for adolescent girls with internalizing problems. Cost Eff Resour Alloc. 2013 Feb 20;11(1):4. doi: 10.1186/1478-7547-11-4. PMID 23425608
- See also: The centers goal is to heighten the scientific competence within the Örebro county through stimulation, initiation and support for research and developement projects. — http://prezi.com/a084vyuggb-7/vfc/?auth_key=002e8aaf28aefd71798b0de15694c3fcea7ea57b